CLINICAL TRIAL: NCT01596413
Title: An Open-label, Cross-over, Pharmacokinetic Study to Assess the Safety and Pharmacokinetics of Transdermal Granisetron (Sancuso® Patch) and IV Granisetron in a Pediatric Oncology Population (Aged 6 to 12 Years)
Brief Title: Pharmacokinetics and Safety of Sancuso and IV Granisetron in Pediatrics Aged 6 to 12 Years
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The company currently does not have plans to conduct this study
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 392MD/46/C
Record Dates: First submitted 2012-04-26; First posted 2012-05-11 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy Induced Nausea and Vomiting
Keywords: CINV
MeSH Terms: conditions — Vomiting | interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sancuso Arm (Experimental): Transdermal Patch 34.3mg graniestron per patch, size 52cm2 Dose: 3.1mg/24 hrs
  Interventions: Drug: Sancuso
- IV Granisetron (Active Comparator): Aqueous solution for IV administration
  1 mg/mL ampoules Dose: 0.01mg/kg (maximum 1 mg)
  Interventions: Drug: IV granisetron

INTERVENTIONS:
Drug: Sancuso — granisetron transdermal system
  Arms: Sancuso Arm
Drug: IV granisetron — IV
  Other Names: IV
  Arms: IV Granisetron

SUMMARY:
The purpose of this study is to determine the dosing strategy for adolescents aged 6 to 12 years.

DETAILED DESCRIPTION:
This is an open-label, multi-center, cross-over study in male and female pediatric cancer patients, aged 6 to 12 years of age who are receiving at least 2 cycles of emetogenic chemotherapy requiring 5-HT3 antagonist treatment of up to 5 days duration. The study is designed to evaluate the safety and PK of transdermal granisetron (Sancuso® patch) in a pediatric population (aged 6 to 12 years), using a population PK approach.

ELIGIBILITY:
Inclusion Criteria:

1. 6 to 12 years of age inclusive at screening.
2. Written patient or parental (or appropriate legal representative) IRB approved informed consent as appropriate.
3. Written patient assent (as appropriate).
4. Confirmed malignancy.
5. Scheduled to receive 2 or more cycles* of emetogenic chemotherapy requiring 5-HT3 antagonist treatment.
6. Scheduled to receive one or more consecutive days of 5-HT3 antagonist treatment, per cycle, as CINV prophylaxis.

   * The cycles of chemotherapy must be consecutive (i.e. one followed by the other) but do not have to be the first and second cycle of a line of treatment.

Exclusion Criteria:

1. Hypersensitivities, allergies or contraindications to study medications; intolerance of medical tape or sticking plaster.
2. Clinical or laboratory signs and symptoms of significant cerebral, cardiovascular, respiratory, renal, hepatobiliary, pancreatic or infectious disease, which in the Investigator's judgment may interfere with the study assessment or completion of the study.
3. Patients with a known history or predisposition to cardiac conduction interval abnormalities, including QT Syndrome, or known family history of long QT Syndrome or taking medications that are known to prolong the QT interval.
4. Patients scheduled to have routine surgery during the study duration.
5. Patients with a life expectancy of < 6 months.
6. Scarring or significant skin disease on both upper arms.
7. Female patients who are pregnant or breast-feeding. All post menarche female patients must have a pregnancy test at screening.
8. Patients who are known or thought to be sexually active must use effective birth control.**
9. Administration of other investigational drugs within 30 days preceding the screening visit, except for anticancer treatments.
10. Any conditions associated with non-compliance.

    * Effective birth control includes absolute abstinence or double barrier birth control methods i.e. condom and one of the following: combined oral contraceptive, diaphragm, depot contraceptive injection.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | Up to 7 days
  Analysis of the plasma concentration of Intravenous granisetron vs transdermal granisetron in pediatric patients receiving chemotherapy over two sequential cycles.

SECONDARY OUTCOMES:
Number of participants with adverse events, application site assessment and clinically significant changes in laboratory assessments over 2 cycles of chemotherapy | From screening until 15 days after the last dose of IV granisetron
  Incidence, frequency, and severity of AEs and SAEs, including clinically significant changes in laboratory assessments and application site assessment.
Number of participants with change in physical assessment including height, weight, BMI and BSA | Through study completion, an average of 8 weeks
  Change in height and weight to calculate BMI and BSA
Number of participants with change in vital signs | Through study completion, an average of 8 weeks
  Change in pulse, systolic and diastolic blood pressures measurements
Number of participants with change in ECG parameters | Through study completion, an average of 8 weeks
  12 lead ECGs will be conducted to time match PK samples after at least 5 minutes supine rest